CLINICAL TRIAL: NCT05188547
Title: Information Retention After Video (Augmented) Preoperative Anesthesiological Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Health Holland (Other); NovaCair (Unknown)
Responsible Party: Principal Investigator, Jan-Wiebe Korstanje, Principle investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MEC-2021-0769
Record Dates: First submitted 2021-12-07; First posted 2022-01-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia; Education; Informed Consent; Anxiety; Multimedia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No video education, only consultation by the anesthesiologist. No knowledge test before the consultation.
- Baseline (No Intervention): No video education, only consultation by the anesthesiologist. Also a knowledge test before the consultation.
- Video (Experimental): Video education and a knowledge test directly afterwards. Consultation by the anesthesiologist after the knowledge test.
  Interventions: Device: Video education
- Video Augmented (Experimental): Video education and consultation by the anesthesiologist directly afterwards. The knowledge test is taken after the consultation.
  Interventions: Device: Video education

INTERVENTIONS:
Device: Video education — Participants will be shown a video educating them on anesthesia and perioperative instructions.
  Arms: Video; Video Augmented

SUMMARY:
Patient education is continuously becoming more important to enable patients to participate in making decisions regarding their medical treatment. Specifically, this is also the case for preoperative education on anesthesia. Worldwide, there are many initiatives to improve preoperative patient education and subsequent level of knowledge of anesthesia, for example by using digital aids. The demand for such aids has increased significantly since the start of the Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) pandemic to facilitate remote preoperative anesthesiological screening. Although many videos to educate patients on anesthesia have been developed and circulate on the internet, there has been little effort to compare this method of educating patients with the traditional one-on-one conversation between the anesthesiologist and the patient.

Objective: To compare short, mid-and long term retention of knowledge after education on anesthesia by watching a video to the traditional one-on-one explanation by the anaesthesiologist.

DETAILED DESCRIPTION:
Participants will be randomized into 4 arms. A control group that will only take the knowledge test after the consultation by the anesthesiologist, a baseline group that will take the knowledge test before and after the consultation to investigate the added value of a knowledge test to knowledge retention. The intervention group is divided into 2 groups. One group will see the educational video and take a knowledge test afterwards. The other group will see the educational video and visit the anesthesiologist afterwards and take the knowledge test after the consultation.

After 2 and 6 weeks patients will be asked to take the knowledge test again, to investigate knowledge retention.

The knowledge test that will be used is the Rotterdam Anesthesia Knowledge Questionnaire currently under development in the Erasmus MC Rotterdam.

ELIGIBILITY:
Inclusion Criteria:

* adults visiting the preoperative anesthesia clinic
* elective surgery
* able to read, write and understand the Dutch language

Exclusion Criteria:

* cardiothoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Information retention short-term | Immediately after the information is provided
  Score on the Rotterdam Anesthesia Knowledge Questionnaire (RAKQ). Results will be expressed as the percentage correct answers of the total number of questions. A higher score means a better knowledge level.

SECONDARY OUTCOMES:
Information retention mid-term | Two weeks after the information is provided compared to directly after the information is provided.
  Difference in score on the Rotterdam Anesthesia Knowledge Questionnaire (RAKQ). Results will be expressed as the percentage correct answers of the total number of questions. A higher score means a better knowledge level.
Anxiety | Immediately after the information is provided
  Difference in score on the APAIS (Amsterdam Preoperative Anxiety and Information Scale). Scores can be between 6 and 30 points, with a higher score meaning a more anxious patient, more in need for information about the surgery and anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Wiebe Korstanje, MD MSc PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol
Time Frame: Within one year after publication, for at least five years
Access Criteria: Whom: Investigators whose proposed use of the data has been approved by the principal investigator or its research team.
  What types of analyses: To achieve aims in the approved proposal What mechanism: Proposals can be filed at our website: https://www.digica-erasmusmc.nl. To gain access requestors will need to sign a data access agreement, data transfer agreement and any other agreement deemed necessary by our institution for safe data sharing.

REFERENCES:
- [Derived] van den Heuvel SF, Jonker P, Hoeks SE, Ismail SY, Stolker RJ, Korstanje JH. The effect of stand-alone and additional preoperative video education on patients' knowledge of anaesthesia: A randomised controlled trial. Eur J Anaesthesiol. 2025 Apr 1;42(4):313-323. doi: 10.1097/EJA.0000000000002109. Epub 2024 Dec 19. PMID 39704038